CLINICAL TRIAL: NCT04901247
Title: Exploring Single Step Culture Medium Refreshment Effect on Embryo Ploidy Rate: A Time-lapse Monitoring Prospective Study
Brief Title: A Time-lapse Monitoring Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Ibrahim Elkhatib, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2103-ABU-003-IK
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Aneuploidy; Infertility
Keywords: infertility; ivf; embryo; embryoscope; culture media; aneuploidy
MeSH Terms: conditions — Aneuploidy; Infertility; Long Qt Syndrome 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- day 3: embryo grading and culture refreshment will be done 67-69 hours post insemination
  Interventions: Behavioral: media refreshment; Behavioral: embryo grading
- day 5: embryo grading and culture medium refreshment will be done 114-118 hours post insemination
  Interventions: Behavioral: media refreshment; Behavioral: embryo grading

INTERVENTIONS:
Behavioral: media refreshment — 20µL of culture medium is aspirated using Eppendorf PCR tips, and freshly, overnight equilibrated 20µL global total LP will be added to the same well
Behavioral: embryo grading — embryo grading should be done prior to media refreshment

SUMMARY:
While numerous types of commercially available human embryo culture media exist for human blastocyst culture, the impact of culture conditions on blastocyst development and aneuploidy formation is not fully understood. Culture conditions are very important for the success of the in vitro fertilization (IVF) cycle, many of the factors involved in the process have been extensively studied. However, none of the studies investigated the effect on euploid rate in a sibling oocyte design with preimplantation genetic testing for aneuploidy (PGT-A), which requires culture till day 7. In addition, the clinical outcome (implantation) will be investigated in a frozen cycle regimen. Hence, the study will explore which day of media refreshment will result in higher rate of ploidy and would improve clinical outcomes. Investigators aim at exploring the best practice, that would empower the euploid rate through the comparison of refreshing the single-step medium on day 3 or day 5 in a sibling oocyte prospective design.

DETAILED DESCRIPTION:
The use of extended embryo culture to the blastocyst stage and PGT-A has enabled identification and selection of embryos with the best developmental potential and improved IVF clinical outcomes. It is considered a routine practice to grade the embryos on day 3 of development, which will require disturbing the culture conditions by annotating the embryos using inverted microscopes. However, the application of Time-lapse technology (TLS) allows annotating the embryos on day 3 without interrupting the culture conditions, especially if TLS is combined with single-step culture medium.

There are several culture factors that can affect embryo development, such as the pH, which is controlled through the concentration of CO2, and also the osmolality, which is the concentration of solute per liter of solution. Evaporation of the solution due to the exposure to high temperature (37°C) can change the concentrations and hence compromise embryo development.

Since single-step medium is designed to sustain embryo development for 5 continuous culture days, while some laboratories culture embryos for 7 days, refreshing the culture medium is inevitable either on day 3 or day 5 of development.

There is no concrete evidence on which of these practices will provide a better environment for embryo development. Moreover, none of the studies investigated the effect of single-step culture medium changeover on day 3 or day 5, on the chromosomal errors (aneuploidy). We aim in this study to explore which day of culture medium refreshment (day 3 or day 5) provides a higher rate of euploid blastocysts.

Summary about data collected. Categorical data will be presented in frequency tables and histograms. Continuous values will be summarized according the mean, standard deviation and confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a minimum of 8 - 10 follicles during ovarian stimulation
* Patients with a minimum of 8 mature oocytes
* PGT-A
* ICSI
* BMI<35
* Age 18- 40
* Fresh or frozen ejaculatory sperm >10,000 motile sperm
* Any Ovarian stimulation
* Embryos cultured in Time-lapse system

Exclusion Criteria:

* PGT-M or PGT-SR
* Previous history of embryo arrest
* Endometriosis
* Hydrosalpinx
* History of uterine abnormality or previous uterine surgery
* History of previous treatment which may impact the ovarian reserve (adnexal surgery, chemotherapy, radiation…)

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Patients undergoing a fertility treatment due to primary or secondary infertility at ART Fertility Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
blastocyst ploidy | 3 days
  determined after biopsy of trophectoderm cells, taken from the blastocyst on day 5, 6 or 7 from development.

SECONDARY OUTCOMES:
cycle ploidy rate | 1 day
  the number of euploid embryos in the group divided by the total number of 2PN
mosaicism frequency | 1 day
  defined as the rate of mosaic errors in aneuploid embryos. This includes full mosaic embryos or aneuploid embryos with 1 or more mosaic chromosome aberration
blastocyst quality at time of biopsy | 1 day
  Four Embryo Quality Scores (EQ1, 2, 3, 4) based on the expansion stage of the blastocyst, the grade of the inner cell mass and the grade of the trophectoderm
blastulation rate | 5 days
  ability of the embryo to form a cavity (=to blastulate) 118hours post ICSI. Number of blastocysts divided by the number of 2PN

CONTACTS AND LOCATIONS:
Overall Officials: IBRAHIM ELKHATIB, Principal Investigator — ART Fertility Clinics LLC
Locations (2):
- United Arab Emirates (2):
  - ART Fertility Clinics, Abu Dhabi
  - Ibrahim Elkhatib, Abu Dhabi

REFERENCES:
- [Background] Bavister BD, Poole KA. Duration and temperature of culture medium equilibration affect frequency of blastocyst development. Reprod Biomed Online. 2005 Jan;10(1):124-9. doi: 10.1016/s1472-6483(10)60813-9. PMID 15705308
- [Background] Costa-Borges N, Belles M, Meseguer M, Galliano D, Ballesteros A, Calderon G. Blastocyst development in single medium with or without renewal on day 3: a prospective cohort study on sibling donor oocytes in a time-lapse incubator. Fertil Steril. 2016 Mar;105(3):707-713. doi: 10.1016/j.fertnstert.2015.11.038. Epub 2015 Dec 12. PMID 26690010
- [Background] Krasnopolskaya KV, Beketova AN, Sesina NI, capital ES, Cyrillichinchenko NK, Badalyan GV, Sudarikova NM, Bocharova TV, Zakharchenko EO. The effect of short-term disturbance of day 3 embryo culture on the development and implantation. Gynecol Endocrinol. 2019;35(sup1):1-4. doi: 10.1080/09513590.2019.1632083. PMID 31532309